CLINICAL TRIAL: NCT04770272
Title: An Adaptive Randomized Neoadjuvant Two Arm Trial in Triple-negative Breast Cancer Comparing a Mono Atezolizumab Window Followed by a Atezolizumab - CTX Therapy With Atezolizumab - CTX Therapy (neoMono)
Brief Title: Study to Compare a Mono Atezolizumab Window Followed by a Atezolizumab - CTX Therapy With Atezolizumab - CTX Therapy
Acronym: neoMono
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial stopped recruitment prematurely after a first planned interim analysis of the first 100 pCR results (given that a probability of less than 2.5% of meeting the primary endpoint was estimated).
Sponsor: Palleos Healthcare GmbH (Industry)
Collaborators: Roche Pharma AG (Industry); Phaon Scientific GmbH (Unknown); University Hospital, Essen (Other); University Hospital Erlangen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Phaon1
Record Dates: First submitted 2021-02-18; First posted 2021-02-25 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Triple-negative Breast Cancer
Keywords: TNBC; Immunotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; Injections; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; Epirubicin; Cyclophosphamide; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): 2 weeks Atezolizumab monotherapy before biopsy, followed by a 12-week therapy with Paclitaxel + Carboplatin+ Atezolizumab every 3 weeks for 4 cycles. This will be followed by Epirubicin + Cyclophosphamide + Atezolizumab every 3 weeks for 4 cycles.
  Interventions: Drug: Atezolizumab 840 MG in 14 ML Injection; Drug: Atezolizumab 1200 MG in 20 ML Injection; Drug: Carboplatin; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide; Procedure: Biopsy Arm A; Procedure: Surgery
- Arm B (Active Comparator): 12-week therapy with Paclitaxel + Carboplatin + Atezolizumab every 3 weeks for 4 cycles. This will be followed by Epirubicin + Cyclophosphamide + Atezolizumab every 3 weeks for 4 cycles.
  Interventions: Drug: Atezolizumab 1200 MG in 20 ML Injection; Drug: Carboplatin; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide; Procedure: Biopsy Arm B; Procedure: Surgery

INTERVENTIONS:
Drug: Atezolizumab 840 MG in 14 ML Injection — 840 mg Day 1 for two weeks
  Other Names: Tecentriq
  Arms: Arm A
Drug: Atezolizumab 1200 MG in 20 ML Injection — 1200 mg Day 1 every 3 weeks for 8 cycles
  Other Names: Tecentriq
Drug: Carboplatin — Dosing according to Area Under the Curve of 2 Intravenous weekly x 12 cycles
  Other Names: Paraplatin
Drug: Paclitaxel — Paclitaxel 80 mg/m² IV weekly x 12 cycles
  Other Names: Abraxane; Onxol
Drug: Epirubicin — 90 mg/m2, day 1 for 4 cycles (12 weeks)
  Other Names: Paxene
Drug: Cyclophosphamide — 600 mg/m2, day 1 for 4 cycles (12 weeks)
  Other Names: Cytoxan
Procedure: Biopsy Arm A — 1st Biopsy two weeks after Baseline visit. 2nd Biopsy after two weeks of Carboplatin + Paclitaxel + Atezolizumab therapy. 3rd Biopsy with tumor size greater 10 mm in diameter.
  Arms: Arm A
Procedure: Biopsy Arm B — 1st Biopsy after two weeks of Carboplatin + Paclitaxel + Atezolizumab therapy. 2nd Biopsy with tumor size greater 10mm in diameter.
  Arms: Arm B
Procedure: Surgery — After completion of 27-28 weeks (Arm B) or 29-30 weeks (Arm A) of neoadjuvant treatment, surgery is planned for all patients.

SUMMARY:
This is a randomized, open-label, adaptive, two arm, multicentre, Phase II trial comparing a neoadjuvant chemotherapy with PDL1-inhibition (Atezolizumab) and Atezolizumab two-week window to chemotherapy with PDL1-inhibition (Atezolizumab) and identify biomarkers predicting (early) response to or resistance against Atezolizumab (alone and with CTX) allowing patients stratification in future clinical trials

DETAILED DESCRIPTION:
This is a randomized, open-label, adaptive, two arm, multicenter phase II trial that enrolled female and male patients with primary TNBC (defined as ER/PR < 10% and HER2-negative) with tumor stages cT1c - cT4d (cN0 and cN+). Patients are randomized to Arm A and B. Randomization is stratified by PD-L1 expression on immune cells (IC-status) and anatomic tumor stage (according to the AJCC 8th edition Anatomic Stage Groups I, II andIII). PD-L1 status is determined by central pathology using the VENTANA PD-L1 (SP142) assay and is defined by PD-L1 IC expression.

Patients in Arm A receive a 2-week monotherapy of Atezolizumab 840 mg q2w prior to initiation of a 12-week neoadjuvant CTX therapy with Paclitaxel 80 mg/m2 i.v. q1w x 12 doses + Carboplatin AUC of 2 i.v. q1w x 12 doses + Atezolizumab 1200 mg day 1 every 3 weeks for 4 doses followed by Epirubicin 90 mg/m2 + Cyclophosphamide 600 mg/m2, both q3w for 4 cycles + Atezolizumab 1200 mg day 1 every 3 weeks for 4 doses.

Patients in Arm B are treated with a neoadjuvant 12-week regimen of Paclitaxel 80 mg/m² i.v. q1w x 12 doses + Carboplatin AUC of 2 i.v. q1w x 12 doses + Atezolizumab 1200 mg day 1 every 3 weeks for 4 doses without a monotherapy window. This is followed by Epirubicin 90 mg/m² + Cyclophosphamide 600 mg/m2, both q3w for 4 cycles + Atezolizumab 1200 mg day 1 every 3 weeks for 4 doses.

Patients in both arms undergo surgery after 29 - 30 weeks therapy in total for Arm A and 27 - 28 weeks therapy in total for Arm B (3 - 4 weeks after last dose of neoadjuvant therapy).

Safety and toxicities under therapy are supervised via regular DSMB meetings. After surgery, patients are treated according to the local SoC therapy for TNBC and followed-up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, age at diagnosis 18 years and above
* Written informed consent prior to admission to this study
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Clinical T1c - T4d
* Stage N0-N3 until 21 patients (5%) with stage N3 are randomized, thereafter N0-N2
* Triple negative breast cancer defined by and confirmed by central pathology:

  * ER negative (<10% positive cells in IHC) and PR negative (<10% positive cells on IHC)
  * HER2 negative breast cancer:

    * Either defined by IHC: ICH scores of 0-1 or an ICH score of 2 in combination with a negative in-situ-hybridization (ISH)
    * Or defined by ISH: negative ISH
* Identifiable PD-L1 IC-status by central pathology (positive or negative) by means of VENTANA PD-L1 (SP142) assay; positive status is defined by PD-L1 expression on IC on ≥ 1% of the tumor area, negative status is defined by PD-L1 expression on IC on < 1% of the tumor area
* No clinical evidence for distant metastasis (cM0)
* Tumor block available for translational research
* Performance Status Eastern Cooperative Oncology Group (ECOG) ≤ 1 or KI ≥ 80 %
* Negative pregnancy test (urine or serum) within 7 days prior to screening in premenopausal patients
* Women of childbearing potential and male patients with partners of childbearing potential must accept to implement a highly effective (less than 1% failure rate according to Pearl index) including at least one non-hormonal contraceptive measures during the study treatment and for 5 months following the last dose of study treatment such as:

  * Intrauterine device (IUD)
  * bilateral tubal occlusion
  * vasectomized partner
  * sexual abstinence
* The patient must be accessible for treatment and follow-up
* Normal cardiac function:

  * Normal electrocardiogram (ECG) (within 6 weeks prior to screening)
  * Normal left ventricular ejection fraction (LVEF) on echocardiorgraphy
* Normal thyroid function

  o Normal TSH and FT4
* Blood counts within 14 days prior screening:

  * absolute neutrophile count (ANC) must be ≥ 1,500/mm3
  * Platelet count must be ≥ 100,000 / mm3
  * Hemoglobin must be ≥ 10 g/dl
* Hepatic functions:

  * Total bilirubin must be ≤ 1 upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation > 1 x ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin
  * Alkaline phosphatase must be ≤ 2.5 x ULN for the lab
  * AST and ALT must be ≤1.5 x ULN for the lab.
  * Patients with AST and ALT or alkaline phosphatase > 1 x ULN are eligible for inclusion if liver imaging (computerized tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET-CT, or PET scan) performed within 3 months prior to randomization (and part of standard of care) does not demonstrate metastatic disease and the requirements in criterion (just above) are met
  * Patients with alkaline phosphatase that is > 1 x ULN but less than or equal to 2.5 x ULN or with unexplained bone pain are eligible if bone imaging does not demonstrate metastatic disease.
  * Creatinine clearance ≥ 40 ml/min performed 28 days prior to screening

Exclusion Criteria:

* Previous history of malign diseases, non-melanoma skin cancer and carcinoma of the cervix are allowed if treated with curative intent
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of Paclitaxel, Carboplatin, Epirubicin, Cyclophosphamide or Atezolizumab
* Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol
* Concurrent treatment with other drugs that are contraindicating the use of the study drugs
* Existing pregnancy
* Breastfeeding
* Sequential breast cancer
* Concurrent treatment with other experimental drugs and participation in another clinical trial or clinical research project (except registry study) within 30 days prior to study entry
* Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study including but not confined to:

  * Uncompensated chronic heart failure or systolic dysfunction (LVEF < 55%, congestive heart failure (CHF) New York Heart Association (NYHA) classes II-IV),
  * unstable arrhythmias requiring treatment i.e., atrial tachycardia with a heart rate ≥ 100/bpm at rest, significant ventricular arrhythmia (ventricular tachycardia) or higher grade AV-block,
  * Angina pectoris within the last 6 months requiring anti-anginal medication,
  * Clinically significant valvular heart disease,
  * Evidence of myocardial infarction on electrocardiogram (ECG),
  * Poorly controlled hypertension (e.g., systolic > 180 mmHg or diastolic > 100 mmHg).
* Inadequate organ function including but not confined to:

  * hepatic impairment as defined by bilirubin > 1.5 x ULN
  * pulmonary disease (severe dyspnea at rest requiring oxygen therapy)
* Abnormal blood values:

  * Platelet count below 100,000/mm3
  * AST/ALT > 1.5 x ULN
  * Hypokalaemia > CTCAE grade 1
  * Neutropenia > CTCAE grade 1
  * Anaemia > CTCAE grade 1
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1 day 1 or anticipation that such a vaccine will be required during the study
* Treatment with systemic immunosuppressive medications (including but not limited to interferons, IL-2) within 28 days or 5 half-lives of the drug, whichever is longer, prior to randomization.
* Treatment with systemic immunosuppressive medications (including but not limited to Prednisone, Cyclophosphamide, Azathioprine, Methotrexate, Thalidomide, and anti-tumor necrosis [anti-TNF] factor agents) within 14 days prior to screening or anticipation of need for systemic immunosuppressive medications during the study
* Patients with prior allogeneic stem cell or solid organ transplantation
* Active or history of autoimmune disease or immune deficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
  * Patients with controlled Type 1 diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are permitted provided all of following conditions are met: Rash must cover < 10% of body surface area; Disease is well controlled at baseline and requires only low-potency topical corticosteroids; No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, Methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral Corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* History of HIV infection, hepatitis B or hepatitis C infection.
* Patients with significant cardiovascular disease
* Patients with inadequate hematological and end-organ function
* Patients receiving therapeutic anti-coagulants
* Stage N3, as soon as 21 patients with stage N3 are randomized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Reiser, Dr., Study Director — Palleos Healthcare GmbH; Hans-Christian Kolberg, Prof. Dr., Principal Investigator — Marienhospital Bottrop gGmbH; Klinik für Frauenheilkunde und Geburtshilfe; 46236 Bottrop
Locations (1):
- Marienhospital Bottrop gGmbH; Klinik für Frauenheilkunde und Geburtshilfe;, Bottrop, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alme AK, Karir BS, Faltas BM, Drake CG. Blocking immune checkpoints in prostate, kidney, and urothelial cancer: An overview. Urol Oncol. 2016 Apr;34(4):171-81. doi: 10.1016/j.urolonc.2016.01.006. Epub 2016 Feb 28. PMID 26923782
- [Background] Bauer KR, Brown M, Cress RD, Parise CA, Caggiano V. Descriptive analysis of estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and HER2-negative invasive breast cancer, the so-called triple-negative phenotype: a population-based study from the California cancer Registry. Cancer. 2007 May 1;109(9):1721-8. doi: 10.1002/cncr.22618. PMID 17387718
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Crittenden M, Kohrt H, Levy R, Jones J, Camphausen K, Dicker A, Demaria S, Formenti S. Current clinical trials testing combinations of immunotherapy and radiation. Semin Radiat Oncol. 2015 Jan;25(1):54-64. doi: 10.1016/j.semradonc.2014.07.003. PMID 25481267
- [Background] Dent R, Trudeau M, Pritchard KI, Hanna WM, Kahn HK, Sawka CA, Lickley LA, Rawlinson E, Sun P, Narod SA. Triple-negative breast cancer: clinical features and patterns of recurrence. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4429-34. doi: 10.1158/1078-0432.CCR-06-3045. PMID 17671126
- [Background] Deyarmin B, Kane JL, Valente AL, van Laar R, Gallagher C, Shriver CD, Ellsworth RE. Effect of ASCO/CAP guidelines for determining ER status on molecular subtype. Ann Surg Oncol. 2013 Jan;20(1):87-93. doi: 10.1245/s10434-012-2588-8. Epub 2012 Aug 9. PMID 22875649
- [Background] Ditsch N, Untch M, Thill M, Muller V, Janni W, Albert US, Bauerfeind I, Blohmer J, Budach W, Dall P, Diel I, Fasching PA, Fehm T, Friedrich M, Gerber B, Hanf V, Harbeck N, Huober J, Jackisch C, Kolberg-Liedtke C, Kreipe HH, Krug D, Kuhn T, Kummel S, Loibl S, Luftner D, Lux MP, Maass N, Mobus V, Muller-Schimpfle M, Mundhenke C, Nitz U, Rhiem K, Rody A, Schmidt M, Schneeweiss A, Schutz F, Sinn HP, Solbach C, Solomayer EF, Stickeler E, Thomssen C, Wenz F, Witzel I, Wockel A. AGO Recommendations for the Diagnosis and Treatment of Patients with Early Breast Cancer: Update 2019. Breast Care (Basel). 2019 Aug;14(4):224-245. doi: 10.1159/000501000. Epub 2019 Aug 6. No abstract available. PMID 31558897
- [Background] Dixon JM, Cameron DA, Arthur LM, Axelrod DM, Renshaw L, Thomas JS, Turnbull A, Young O, Loman CA, Jakubowski D, Baehner FL, Singh B. Accurate Estrogen Receptor Quantification in Patients with Negative and Low-Positive Estrogen-Receptor-Expressing Breast Tumors: Sub-Analyses of Data from Two Clinical Studies. Adv Ther. 2019 Apr;36(4):828-841. doi: 10.1007/s12325-019-0896-0. Epub 2019 Mar 11. PMID 30859501
- [Background] Dowsett M, Smith IE, Ebbs SR, Dixon JM, Skene A, Griffith C, Boeddinghaus I, Salter J, Detre S, Hills M, Ashley S, Francis S, Walsh G; IMPACT Trialists. Short-term changes in Ki-67 during neoadjuvant treatment of primary breast cancer with anastrozole or tamoxifen alone or combined correlate with recurrence-free survival. Clin Cancer Res. 2005 Jan 15;11(2 Pt 2):951s-8s. PMID 15701892
- [Background] Dowsett M, Smith I, Robertson J, Robison L, Pinhel I, Johnson L, Salter J, Dunbier A, Anderson H, Ghazoui Z, Skene T, Evans A, A'Hern R, Iskender A, Wilcox M, Bliss J. Endocrine therapy, new biologicals, and new study designs for presurgical studies in breast cancer. J Natl Cancer Inst Monogr. 2011;2011(43):120-3. doi: 10.1093/jncimonographs/lgr034. PMID 22043057
- [Background] Gelman A, Stern HS, Carlin JB, Dunson DB, Vehtari A & Rubin DB. Bayesian data analysis. Chapman and Hall/CRC. 2013
- [Background] Gianni L, Huang CS, Egle D, Bermejo B, Zamagni C & Thill M (2019, Dezember 12). Combining Atezolizumab with Neoadjuvant Chemotherapy Does Not Improve Pathologic Complete Response Rates for Patients with Triple-Negative Breast Cancer. SABCS 2019, Marc.
- [Background] Gluz O, Liedtke C, Gottschalk N, Pusztai L, Nitz U, Harbeck N. Triple-negative breast cancer--current status and future directions. Ann Oncol. 2009 Dec;20(12):1913-27. doi: 10.1093/annonc/mdp492. Epub 2009 Nov 9. PMID 19901010
- [Background] Gluz O, Kolberg-Liedtke C, Prat A, Christgen M, Gebauer D, Kates R, Pare L, Grischke EM, Forstbauer H, Braun M, Warm M, Hackmann J, Uleer C, Aktas B, Schumacher C, Kuemmel S, Wuerstlein R, Pelz E, Nitz U, Kreipe HH, Harbeck N. Efficacy of deescalated chemotherapy according to PAM50 subtypes, immune and proliferation genes in triple-negative early breast cancer: Primary translational analysis of the WSG-ADAPT-TN trial. Int J Cancer. 2020 Jan 1;146(1):262-271. doi: 10.1002/ijc.32488. Epub 2019 Jun 19. PMID 31162838
- [Background] Gluz O, Nitz U, Liedtke C, Christgen M, Grischke EM, Forstbauer H, Braun M, Warm M, Hackmann J, Uleer C, Aktas B, Schumacher C, Bangemann N, Lindner C, Kuemmel S, Clemens M, Potenberg J, Staib P, Kohls A, von Schumann R, Kates R, Kates R, Schumacher J, Wuerstlein R, Kreipe HH, Harbeck N. Comparison of Neoadjuvant Nab-Paclitaxel+Carboplatin vs Nab-Paclitaxel+Gemcitabine in Triple-Negative Breast Cancer: Randomized WSG-ADAPT-TN Trial Results. J Natl Cancer Inst. 2018 Jun 1;110(6):628-637. doi: 10.1093/jnci/djx258. PMID 29228315
- [Background] Houssami N, Macaskill P, von Minckwitz G, Marinovich ML, Mamounas E. Meta-analysis of the association of breast cancer subtype and pathologic complete response to neoadjuvant chemotherapy. Eur J Cancer. 2012 Dec;48(18):3342-54. doi: 10.1016/j.ejca.2012.05.023. Epub 2012 Jul 3. PMID 22766518
- [Background] Ibrahim JG, Chen MH & Sinha, D. (2014). Bayesian Survival Analysis. In N. Balakrishnan, T. Colton, B. Everitt, W. Piegorsch, F. Ruggeri, & J. L. Teugels (Hrsg.), Wiley StatsRef: Statistics Reference Online (S. stat06003). John Wiley & Sons
- [Background] Iwamoto T, Booser D, Valero V, Murray JL, Koenig K, Esteva FJ, Ueno NT, Zhang J, Shi W, Qi Y, Matsuoka J, Yang EJ, Hortobagyi GN, Hatzis C, Symmans WF, Pusztai L. Estrogen receptor (ER) mRNA and ER-related gene expression in breast cancers that are 1% to 10% ER-positive by immunohistochemistry. J Clin Oncol. 2012 Mar 1;30(7):729-34. doi: 10.1200/JCO.2011.36.2574. Epub 2012 Jan 30. PMID 22291085
- [Background] Keup C, Storbeck M, Hauch S, Hahn P, Sprenger-Haussels M, Tewes M, Mach P, Hoffmann O, Kimmig R, Kasimir-Bauer S. Cell-Free DNA Variant Sequencing Using CTC-Depleted Blood for Comprehensive Liquid Biopsy Testing in Metastatic Breast Cancer. Cancers (Basel). 2019 Feb 18;11(2):238. doi: 10.3390/cancers11020238. PMID 30781720
- [Background] Klein JP & Moeschberger ML (2010). Survival analysis: Techniques for censored and truncated data (2. ed., corr. 3. print). Springer.
- [Background] Lee HJ, Lee JJ, Song IH, Park IA, Kang J, Yu JH, Ahn JH, Gong G. Prognostic and predictive value of NanoString-based immune-related gene signatures in a neoadjuvant setting of triple-negative breast cancer: relationship to tumor-infiltrating lymphocytes. Breast Cancer Res Treat. 2015 Jun;151(3):619-27. doi: 10.1007/s10549-015-3438-8. Epub 2015 May 26. PMID 26006068
- [Background] Kolberg-Liedtke C, Feuerhake F, Garke M, Christgen M, Kates R, Grischke EM, Forstbauer H, Braun M, Warm M, Hackmann J, Uleer C, Aktas B, Schumacher C, Kuemmel S, Wuerstlein R, Graeser M, Nitz U, Kreipe H, Gluz O, Harbeck N. Impact of stromal tumor-infiltrating lymphocytes (sTILs) on response to neoadjuvant chemotherapy in triple-negative early breast cancer in the WSG-ADAPT TN trial. Breast Cancer Res. 2022 Sep 2;24(1):58. doi: 10.1186/s13058-022-01552-w. PMID 36056374
- [Background] Liedtke C, Mazouni C, Hess KR, Andre F, Tordai A, Mejia JA, Symmans WF, Gonzalez-Angulo AM, Hennessy B, Green M, Cristofanilli M, Hortobagyi GN, Pusztai L. Response to neoadjuvant therapy and long-term survival in patients with triple-negative breast cancer. J Clin Oncol. 2008 Mar 10;26(8):1275-81. doi: 10.1200/JCO.2007.14.4147. Epub 2008 Feb 4. PMID 18250347
- [Background] Llombart-Cussac A, Cortes J, Pare L, Galvan P, Bermejo B, Martinez N, Vidal M, Pernas S, Lopez R, Munoz M, Nuciforo P, Morales S, Oliveira M, de la Pena L, Pelaez A, Prat A. HER2-enriched subtype as a predictor of pathological complete response following trastuzumab and lapatinib without chemotherapy in early-stage HER2-positive breast cancer (PAMELA): an open-label, single-group, multicentre, phase 2 trial. Lancet Oncol. 2017 Apr;18(4):545-554. doi: 10.1016/S1470-2045(17)30021-9. Epub 2017 Feb 24. PMID 28238593
- [Background] Loi S, Schmid P, Aktan G, Karantza V & Salgado R (2019). 4O Relationship between tumor infiltrating lymphocytes (TILs) and response to pembrolizumab (pembro)+ chemotherapy (CT) as neoadjuvant treatment (NAT) for triple-negative breast cancer (TNBC): Phase Ib KEYNOTE-173 trial. Annals of Oncology
- [Background] Loibl S, Untch M, Burchardi N, Huober J, Sinn BV, Blohmer JU, Grischke EM, Furlanetto J, Tesch H, Hanusch C, Engels K, Rezai M, Jackisch C, Schmitt WD, von Minckwitz G, Thomalla J, Kummel S, Rautenberg B, Fasching PA, Weber K, Rhiem K, Denkert C, Schneeweiss A. A randomised phase II study investigating durvalumab in addition to an anthracycline taxane-based neoadjuvant therapy in early triple-negative breast cancer: clinical results and biomarker analysis of GeparNuevo study. Ann Oncol. 2019 Aug 1;30(8):1279-1288. doi: 10.1093/annonc/mdz158. PMID 31095287
- [Background] Loibl S, Werutsky G, Nekljudova V, Seiler S, Blohmer JU, Denkert C, Hanusch C, Huober JB, Jackisch C, Kummel S, Schneeweiss A, Untch M, Rhiem K, Fasching PA, Von Minckwitz G & Furlanetto J (2017). Impact in delay of start of chemotherapy and surgery on pCR and survival in breast cancer: A pooled analysis of individual patient data from six prospectively randomized neoadjuvant trials. Journal of Clinical Oncology
- [Background] Marra A, Viale G, Curigliano G. Recent advances in triple negative breast cancer: the immunotherapy era. BMC Med. 2019 May 9;17(1):90. doi: 10.1186/s12916-019-1326-5. PMID 31068190
- [Background] Matsushita M, Kawaguchi M. Immunomodulatory Effects of Drugs for Effective Cancer Immunotherapy. J Oncol. 2018 Oct 25;2018:8653489. doi: 10.1155/2018/8653489. eCollection 2018. PMID 30498512
- [Background] Foulds GA, Vadakekolathu J, Abdel-Fatah TMA, Nagarajan D, Reeder S, Johnson C, Hood S, Moseley PM, Chan SYT, Pockley AG, Rutella S, McArdle SEB. Immune-Phenotyping and Transcriptomic Profiling of Peripheral Blood Mononuclear Cells From Patients With Breast Cancer: Identification of a 3 Gene Signature Which Predicts Relapse of Triple Negative Breast Cancer. Front Immunol. 2018 Sep 11;9:2028. doi: 10.3389/fimmu.2018.02028. eCollection 2018. PMID 30254632
- [Background] Nuciforo P, Pascual T, Cortes J, Llombart-Cussac A, Fasani R, Pare L, Oliveira M, Galvan P, Martinez N, Bermejo B, Vidal M, Pernas S, Lopez R, Munoz M, Garau I, Manso L, Alarcon J, Martinez E, Rodrik-Outmezguine V, Brase JC, Villagrasa P, Prat A, Holgado E. A predictive model of pathologic response based on tumor cellularity and tumor-infiltrating lymphocytes (CelTIL) in HER2-positive breast cancer treated with chemo-free dual HER2 blockade. Ann Oncol. 2018 Jan 1;29(1):170-177. doi: 10.1093/annonc/mdx647. PMID 29045543
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Park MM, Ebel JJ, Zhao W, Zynger DL. ER and PR immunohistochemistry and HER2 FISH versus oncotype DX: implications for breast cancer treatment. Breast J. 2014 Jan-Feb;20(1):37-45. doi: 10.1111/tbj.12223. Epub 2013 Nov 22. PMID 24261318
- [Background] Raghav KP, Hernandez-Aya LF, Lei X, Chavez-Macgregor M, Meric-Bernstam F, Buchholz TA, Sahin A, Do KA, Hortobagyi GN, Gonzalez-Angulo AM. Impact of low estrogen/progesterone receptor expression on survival outcomes in breast cancers previously classified as triple negative breast cancers. Cancer. 2012 Mar 15;118(6):1498-506. doi: 10.1002/cncr.26431. Epub 2011 Aug 11. PMID 21837669
- [Background] Raja R, Kuziora M, Brohawn PZ, Higgs BW, Gupta A, Dennis PA, Ranade K. Early Reduction in ctDNA Predicts Survival in Patients with Lung and Bladder Cancer Treated with Durvalumab. Clin Cancer Res. 2018 Dec 15;24(24):6212-6222. doi: 10.1158/1078-0432.CCR-18-0386. Epub 2018 Aug 9. PMID 30093454
- [Background] Royston P & Sauerbrei W (2008). Multivariable Model-Building. John Wiley & Sons, Ltd.
- [Background] Saliou A, Bidard FC, Lantz O, Stern MH, Vincent-Salomon A, Proudhon C, Pierga JY. Circulating tumor DNA for triple-negative breast cancer diagnosis and treatment decisions. Expert Rev Mol Diagn. 2016;16(1):39-50. doi: 10.1586/14737159.2016.1121100. Epub 2015 Dec 9. PMID 26568208
- [Background] Sanford RA, Song J, Gutierrez-Barrera AM, Profato J, Woodson A, Litton JK, Bedrosian I, Albarracin CT, Valero V, Arun B. High incidence of germline BRCA mutation in patients with ER low-positive/PR low-positive/HER-2 neu negative tumors. Cancer. 2015 Oct 1;121(19):3422-7. doi: 10.1002/cncr.29572. Epub 2015 Aug 17. PMID 26280679
- [Background] Schmid P, Cortés J, Dent R, Pusztai L, McArthur HL, Kuemmel S, Bergh J, Denkert C, Park YH & Hui R (2019). KEYNOTE-522: Phase III study of pembrolizumab (pembro)+ chemotherapy (chemo) vs placebo (pbo)+ chemo as neoadjuvant treatment, followed by pembro vs pbo as adjuvant treatment for early triple-negative breast cancer (TNBC). Annals of Oncology
- [Background] Schmid P. ESMO 2018 presidential symposium-IMpassion130: atezolizumab+nab-paclitaxel in triple-negative breast cancer. ESMO Open. 2018 Oct 20;3(6):e000453. doi: 10.1136/esmoopen-2018-000453. eCollection 2018. No abstract available. PMID 30425847
- [Background] Sharma P, Allison JP. The future of immune checkpoint therapy. Science. 2015 Apr 3;348(6230):56-61. doi: 10.1126/science.aaa8172. PMID 25838373
- [Background] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Background] Slovin SF, Higano CS, Hamid O, Tejwani S, Harzstark A, Alumkal JJ, Scher HI, Chin K, Gagnier P, McHenry MB, Beer TM. Ipilimumab alone or in combination with radiotherapy in metastatic castration-resistant prostate cancer: results from an open-label, multicenter phase I/II study. Ann Oncol. 2013 Jul;24(7):1813-1821. doi: 10.1093/annonc/mdt107. Epub 2013 Mar 27. PMID 23535954
- [Background] Sokolenko AP, Imyanitov EN. Molecular Tests for the Choice of Cancer Therapy. Curr Pharm Des. 2017;23(32):4794-4806. doi: 10.2174/1381612823666170719110125. PMID 28721808
- [Background] Sorlie T, Perou CM, Tibshirani R, Aas T, Geisler S, Johnsen H, Hastie T, Eisen MB, van de Rijn M, Jeffrey SS, Thorsen T, Quist H, Matese JC, Brown PO, Botstein D, Lonning PE, Borresen-Dale AL. Gene expression patterns of breast carcinomas distinguish tumor subclasses with clinical implications. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10869-74. doi: 10.1073/pnas.191367098. PMID 11553815
- [Background] Tan W, Yang M, Yang H, Zhou F, Shen W. Predicting the response to neoadjuvant therapy for early-stage breast cancer: tumor-, blood-, and imaging-related biomarkers. Cancer Manag Res. 2018 Oct 9;10:4333-4347. doi: 10.2147/CMAR.S174435. eCollection 2018. PMID 30349367
- [Background] Thompson RH, Dong H, Lohse CM, Leibovich BC, Blute ML, Cheville JC, Kwon ED. PD-1 is expressed by tumor-infiltrating immune cells and is associated with poor outcome for patients with renal cell carcinoma. Clin Cancer Res. 2007 Mar 15;13(6):1757-61. doi: 10.1158/1078-0432.CCR-06-2599. PMID 17363529
- [Background] Tibshirani R (1996). Regression Shrinkage and Selection via the Lasso. Journal of the Royal Statistical Society. Series B (Methodological)
- [Background] Untch M, Jackisch C, Schneeweiss A, Conrad B, Aktas B, Denkert C, Eidtmann H, Wiebringhaus H, Kummel S, Hilfrich J, Warm M, Paepke S, Just M, Hanusch C, Hackmann J, Blohmer JU, Clemens M, Darb-Esfahani S, Schmitt WD, Dan Costa S, Gerber B, Engels K, Nekljudova V, Loibl S, von Minckwitz G; German Breast Group (GBG); Arbeitsgemeinschaft Gynakologische Onkologie-Breast (AGO-B) Investigators. Nab-paclitaxel versus solvent-based paclitaxel in neoadjuvant chemotherapy for early breast cancer (GeparSepto-GBG 69): a randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):345-356. doi: 10.1016/S1470-2045(15)00542-2. Epub 2016 Feb 8. PMID 26869049
- [Background] Yang B, Chou J, Tao Y, Wu D, Wu X, Li X, Li Y, Chu Y, Tang F, Shi Y, Ma L, Zhou T, Kaufmann W, Carey LA, Wu J, Hu Z. An assessment of prognostic immunity markers in breast cancer. NPJ Breast Cancer. 2018 Oct 29;4:35. doi: 10.1038/s41523-018-0088-0. eCollection 2018. PMID 30393759
- [Background] Yi M, Huo L, Koenig KB, Mittendorf EA, Meric-Bernstam F, Kuerer HM, Bedrosian I, Buzdar AU, Symmans WF, Crow JR, Bender M, Shah RR, Hortobagyi GN, Hunt KK. Which threshold for ER positivity? a retrospective study based on 9639 patients. Ann Oncol. 2014 May;25(5):1004-11. doi: 10.1093/annonc/mdu053. Epub 2014 Feb 20. PMID 24562447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at 34 centers in Germany.The expected number of patients to be recruited was 458. As the study protocol mandated termination of trial recruitment based on the results of the first interim analysis, the final Intention-to-treat (ITT) population was limited to 359 participants.442 participants had been screened, and 2 per arm were excluded from analysis due to protocol violations. First participant enrolled: 2021-03-01; last visit of a participant: 2024-10-02.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 180 (2 more had been enrolled, but were subsequently excluded from analysis during the data review meeting due to violation of inclusion/exclusion.) | 179 (2 more had been enrolled, but were subsequently excluded from analysis during the data review meeting due to violation of inclusion/exclusion.)
Completed | 134 | 131
Not Completed | 46 | 48
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 23 | 21
Not completed — Physician Decision | 7 | 3
Not completed — Disease progression | 4 | 8
Not completed — Switched to other therapy. | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 180 | 179 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.57 (11.66) | 49.98 (12.34) | 49.27 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 179 | 358
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 168 | 171 | 339
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  Germany | 180 | 179 | 359
ECOG [Count of Participants; unit: Participants] — ECOG scales (Eastern Cooperative Oncology Group Performance Status) are 0-to-5 rating systems used in oncology to assess a cancer patient's functional ability and overall well-being, helping doctors decide on treatments, predict outcomes, and determine eligibility for clinical trials, with 0 being fully active and 5 being deceased, reflecting a patient's capacity for daily activities, self-care, and work
  Participants
    ECOG = 0 | 169 | 170 | 339
    ECOG = 1 | 11 | 9 | 20
HER2 IHC status [Count of Participants; unit: Participants] — HER2 IHC (Immunohistochemistry) status describes the amount of HER2 protein on cancer cells, scored 0 to 3+; 3+ means HER2-Positive (lots of protein, good for targeted drugs), 0 or 1+ usually means HER2-Negative, and 2+ is Equivocal/Borderline, requiring further testing (like FISH) for confirmation, with newer categories like HER2-Low (1+ or 2+/ISH-negative) now recognized for specific therapies.
  Participants
    0 | 72 | 75 | 147
    1+ | 80 | 82 | 162
    2+ | 28 | 22 | 50
Tumor histology [Count of Participants; unit: Participants] — Breast tumor histology examines cell structure, differentiation, and arrangement (like tubules, nests, or single files) to classify tumors (e.g., ductal, lobular, mucinous, papillary) and grade aggressiveness (e.g., tubule formation, nuclear pleomorphism, mitotic count), revealing key features like invasion of basement membranes (invasive carcinoma) versus confined growth (DCIS), crucial for diagnosis, prognosis, and treatment planning.
  Participants
    INFILTRATING DUCTAL | 171 | 166 | 337
    INFILTRATING LOBULAR | 3 | 0 | 3
    MIXED | 1 | 2 | 3
    MUCINOUS | 0 | 1 | 1
    Missing | 5 | 10 | 15
Tumor grading [Count of Participants; unit: Participants] — Tumor grading is a system that classifies cancer cells based on how abnormal they look under a microscope, indicating their likely behavior (how fast they grow and spread). Grades typically range from 1 to 4, with Grade 1 (well-differentiated) cells resembling normal cells and growing slowly, while Grade 4 (undifferentiated/poorly differentiated) cells look very abnormal, grow aggressively, and spread quickly. This grading helps doctors plan treatment and predict prognosis, working alongside cancer staging (which describes the tumor's size and spread).
  Participants
    GRADE 2 | 21 | 18 | 39
    GRADE 3 | 159 | 161 | 320
Tumor stage [Count of Participants; unit: Participants] — In breast cancer staging, the "cT" refers to the clinical tumor stage, determined by physical exam/imaging (like CT scans), describing the primary tumor's size and local spread (e.g., T1, T2, T3, T4), indicating if it's small, large, or growing into skin/chest wall, a crucial part of the TNM system (Tumor, Nodes, Metastasis) that helps define the cancer's extent before treatment begins.
  Participants
    cT1c | 73 | 63 | 136
    cT2 | 96 | 102 | 198
    cT3 | 6 | 12 | 18
    cT4a | 1 | 0 | 1
    cT4b | 1 | 1 | 2
    cT4c | 1 | 0 | 1
    cT4d | 2 | 1 | 3
Nodal status [Count of Participants; unit: Participants] — Nodal status in breast cancer refers to whether cancer cells have spread to nearby lymph nodes (usually under the arm), a key factor for staging, prognosis, and treatment planning, classified under the TNM system (N0 for no spread, N1-N3 for increasing involvement). It's assessed via sentinel lymph node biopsy or axillary dissection, with positive nodes indicating higher risk, guiding decisions for systemic therapies like chemotherapy, even if the primary tumor seems small.
  Participants
    cN0 | 123 | 126 | 249
    cN1 | 41 | 43 | 84
    cN2 | 10 | 7 | 17
    cN3 | 6 | 3 | 9
HER2 status [Count of Participants; unit: Participants] — HER2 IHC (Immunohistochemistry) status describes the amount of HER2 protein on cancer cells, scored 0 to 3+; 3+ means HER2-Positive (lots of protein, good for targeted drugs), 0 or 1+ usually means HER2-Negative, and 2+ is Equivocal/Borderline, requiring further testing (like FISH) for confirmation, with newer categories like HER2-Low (1+ or 2+/ISH-negative) now recognized for specific therapies.
  Participants
    LOW (IHC 1+ or 2+/ISH negative) | 108 | 104 | 212
    NEGATIVE | 72 | 75 | 147
    POSITIVE | 0 | 0 | 0
Hormone receptor status [Count of Participants; unit: Participants]
  Borderline Positive (either ER or PR expression is above 1% and <10%) | 25 | 33 | 58
  Negative | 155 | 146 | 301
Weight (kg) [Median (Standard Deviation); unit: kg] | 72.00 (13.52) | 70.36 (13.65) | 71.18 (13.60)
Percentage of Positive KI-67 Cells [Mean (Standard Deviation); unit: percentage] — Positive Ki-67 cells are cells actively dividing or preparing to divide, identified by the presence of the Ki-67 protein, a key marker for cell proliferation used in cancer diagnosis to gauge tumor aggressiveness (proliferation index) and predict treatment response, especially in breast cancer, where higher percentages often signal faster-growing tumors, though cutoffs vary.
  percentage | 69.28 (17.97) | 69.26 (17.86) | 69.27 (17.89)
Cellularity (percentage of tumor volume occupied by invasive tumors cells) [Mean (Standard Deviation); unit: percentage] — Cellularity in breast cancer refers to the density or proportion of cancer cells within the tumor, a key factor pathologists assess in tissue samples (H&E slides) to gauge tumor aggressiveness, treatment response (especially after neoadjuvant therapy), and patient prognosis, often linked to tumor size and vascular invasion, with high cellularity sometimes indicating worse outcomes.
  percentage | 39.22 (20.17) | 38.80 (20.88) | 39.01 (20.50)
TILs (percentage) [Mean (Standard Deviation); unit: percentage] — Tumor-infiltrating lymphocytes (TILs) are immune cells found within and around breast cancer tumors. Their presence indicates the body is mounting an anti-tumor immune response and serves as an important prognostic and predictive biomarker, especially in certain breast cancer subtypes, whereby a higher percentage is often associated with a better prognosis.
  percentage | 24.68 (19.64) | 25.10 (19.38) | 24.89 (19.49)
PD-L1 expression [Mean (Standard Deviation); unit: percentage] — PD-L1 expression is primarily measured in tumor tissue samples using immunohistochemistry (IHC), a laboratory technique where pathologists visually assess stained tissue under a microscope. This measurement helps determine if a patient is likely to benefit from immune checkpoint inhibitor therapies (immunotherapy).
  percentage | 1.12 (2.77) | 1.22 (3.55) | 1.17 (3.18)
Largest tumor diameter [Mean (Standard Deviation); unit: mm] | 24.79 (2.47) | 25.34 (11.52) | 25.07 (11.99)

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (ypT0/is, ypN0)
Description: Pathological Complete Response defined as no residual invasive tumor cells in the breast and in the lymph nodes (ypT0/is, ypN0).
Time Frame: after 29-30 weeks in Arm A and after 27-28 weeks in Arm B.
Population: The analysis was performed in the ITT population. The analysis population for the primary endpoint encompassed 339 patients with available pCR status (10 missing in each arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 170 | 169
Participants
  pCR = 0 (no pCR) | 58 | 52
  pCR = 1 (pCR achieved) | 112 | 117
Statistical Analysis 1: Comparison: Arm A vs Arm B; This was a randomized, open-label, adaptive, two arm, multicenter phase II trial that enrolled female and male patients with primary TNBC (defined as ER/PR < 10% and HER2-negative) with tumor stages cT1c - cT4d (cN0 and cN+). Patients were randomized to Arm A and B, stratified by PD-L1 expression on immune cells (IC-status) and anatomic tumor stage (Anatomic Stage Groups I, II and III). PD-L1 status was determined by central pathology using the VENTANA PD-L1 (SP142) assay; Test type: Superiority — The primary analysis uses Bayesian statistics for proportions, and is based on non-informative uniform (beta) priors for the pCR rates pA and pB in arms A (experimental) and B (control) respectively. Similar to a proof-of-concept trial, a dual criterion to simultaneously test for significant and relevant superiority at different levels of certainty was used, by requiring posterior probabilities, conditional on observed response counts xA, xB respectively in the two arms; Risk Difference (RD) = -0.0327, 95% CI 2-sided [-0.1307 to 0.0663]

2. Secondary Outcome: Number of Adverse Events by Grade
Description: Safety (incidence, relationship, seriousness, and severity of all AEs, SAEs, AESIs coded by medical dictionary for regulatory activities (MedDRA), summarized by Preferred Term and System Organ Class and graded according to common terminology criteria of adverse events (CTCAE V5.0)
Time Frame: from date of randomization up to 24 months
Population: Safety endpoints are based on a subset of the ITT population that actually received treatment. The safety population included 356 patients, 178 from Arm A and 178 from Arm B. Most frequent AEs (>10% of patients) by system organ class are shown.
Measure: Number; unit: Adverse Events
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 178 | 178
Adverse Events
  CTCAE grade - all | 3281 | 3313
  CTCAE grade 1 | 1924 | 1937
  CTCAE grade 2 | 847 | 849
  CTCAE grade 3 | 376 | 368
  CTCAE grade 4 | 133 | 159
  CTCAE grade 5 | 1 | 0

3. Secondary Outcome: Pathological Complete Response (ypT0/is, ypN0) (ER/PR Expression of <1%).
Description: Pathological complete response defined as no residual invasive tumor cells in the breast and in the lymph nodes (ypT0/is, ypN0) in patients with an ER/PR expression of <1% and an ER/PR expression of 1% to 10%.
Time Frame: after 29-30 weeks in Arm A and after 27-28 weeks in Arm B
Population: Patients with an ER/PR expression of <1%. (Data for partients and an ER/PR expression of 1% to 10%, see below.)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 147 | 138
Participants
  pCR = 0 (no pCR) | 53 | 44
  pCR = 1 (pCR achieved) | 94 | 94
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.0411, 95% CI 2-sided [-0.1497 to 0.0689]

4. Secondary Outcome: Pathological Complete Response (ypT0/is, ypN0) (ER/PR Between 1 and 10 %).
Description: as for outcome 3
Time Frame: after 29-30 weeks in Arm A and after 27-28 weeks in Arm B
Population: Patients with an ER/PR expression of 1% to 10%. (Data for partients an ER/PR expression of <1%, see above.)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 23 | 31
Participants
  pCR = 0 (no pCR) | 5 | 8
  pCR = 1 (pCR achieved) | 18 | 23
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = 0.0323, 95% CI 2-sided [-0.1957 to 0.2524]

5. Secondary Outcome: Pathological Complete Response (ypT0, ypN0)
Description: Pathological complete response defined as no tumor cells (invasive and no non-invasive) in the breast but also in the lymph nodes (ypN0, ypT0).
Time Frame: after 29-30 weeks in Arm A and after 27-28 weeks in Arm B.
Population: Same as f0r Primary Endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 170 | 169
Participants
  pCR (ypT0, ypN0) = 0 (not achieved) | 67 | 58
  pCR (ypT0, ypN0) = 1 (achieved) | 103 | 111
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.051, 95% CI 2-sided [-0.153 to 0.051]

6. Secondary Outcome: Near Pathological Complete Response (Near pCR)
Description: Near pCR defined as residual tumor <5 mm in the breast irrespective of in situ and lymph nodes status
Time Frame: after 29-30 weeks in Arm A and after 27-28 weeks in Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 170 | 170
Participants
  pCR (ypT0/is/1a) = 0 | 38 | 31
  pCR (ypT0/is/1a) = 1 | 132 | 139
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.041, 95% CI 2-sided [-0.127 to 0.044]

7. Secondary Outcome: Pathological Complete Response (no Invasive Tumor)
Description: Pathological Complete Response defined as no invasive tumor in the breast, irrespective of lymph node status
Time Frame: after 29-30 weeks in Arm A and after 27-28 weeks in Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 170 | 170
Participants
  pCR (ypT0) = 0 | 63 | 52
  pCR (ypT0) = 1 | 107 | 118
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.064, 95% CI 2-sided [-0.166 to 0.034]

8. Secondary Outcome: Decrease of Ki-67 Expression by ≥ 30% Compared to Baseline as Continuous Predictor After 14 (Arm A)/28 Days (armB) (+/- 2 Days) of Treatment
Description: Decrease of Ki-67 expression versus baseline after 14/28 days (+/- 2 days) of treatment as continuous predictor.
  General comment to analysis of secondary biomarker endpoints: biomarker endpoints are analysed as secondary efficacy endpoints. Biomarker endpoints are measured by core biopsy at a central pathology laboratory at two different timepoints. For arm A visit 1 (A1 in tables) corresponds to day 14 in the trial and denotes the measurement after the Atezolizumab monotherapy window. Arm A visit 3 (A3 in tables) corresponds to day 28 and denotes a measurement taken again after two weeks of combined immuno- and chemotherapy. In arm B, only visit 2 (day 14; B2 in tables) is measured after the initial two weeks of combined immuno- and chemotherapy.
Time Frame: after 14/28 days (+/- 2 days) of treatment
Population: Analyzed were available samples of participants (20 missing in arm A; 41 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 160 | 138
Participants
  Ki-67 BL Decr. >= 30% A1B2 = 0 (not achieved) | 142 | 90
  Ki-67 BL Decr. >= 30% A1B2 = 1 (achieved) | 18 | 48
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.233, 95% CI 2-sided [-0.326 to -0.14] — CI given as High posterior density interval (Bayesian confidence interval based on posterior distribution of effect/parameter of interest)

9. Secondary Outcome: Decrease of Ki-67 Expression After 28 Days (+/- 2 Days) of Treatment for Arm A and Arm B.
Description: Decrease of Ki-67 expression versus baseline by 30% or more after 28 days (+/- 2 days) of treatment. See general comments to biomarker endpoints above. Decrease of Ki-67 defined as ≥ 30% compared to baseline.
Time Frame: after 28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (43 missing in arm A; 41 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 137 | 138
Participants
  Ki-67 BL Decr. >= 30% A3B2 = 0 (not achieved) | 84 | 90
  Ki-67 BL Decr. >= 30% A3B2 = 1 (achieved) | 53 | 48
Statistical Analysis 1: Comparison: Arm A; Test type: Superiority; Risk Difference (RD) = 0.039, 95% CI 2-sided [-0.078 to 0.15] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Stromal Tumor-infiltrating Lymphocytes (TILs) ≥ 60% After 14 (Arm A)/28 Days (ArmB)
Description: TILs after 14/28 days (+/- 2 days) of treatment as continuous predictor. See general comments to biomarker endpoints above.
Time Frame: after 14/28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (20 missing in arm A; 39 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 160 | 140
Participants
  TILs >= 60% A1B2 = 0 (not achieved) | 134 | 96
  TILs >= 60% A1B2 = 1 (achieved) | 26 | 44
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.15, 95% CI 2-sided [-0.245 to -0.054] — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: Tumor-infiltrating Lymphocytes (TILs) ≥ 60% After 28 Days
Description: TILs ≥ 60% after 28 days (+/- 2 days) of treatment. Stromal Tumor Infiltrating Lymphocytes (TILs) ≥ 60%.
  See general comments to biomarker endpoints above.
Time Frame: after 28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (42 missing in arm A; 39 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 138 | 140
Participants
  TILs >= 60% A3B2 = 0 (not achieved) | 102 | 96
  TILs >= 60% A3B2 = 1 (achieved) | 36 | 44
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.052, 95% CI 2-sided [-0.157 to 0.055] — [estimate comment as in outcome 8, analysis 1]

12. Secondary Outcome: Complete Cell Cycle Arrest (CCCA) After 14 (Arm A)/28 Days (armB) (+/- 2 Days) of Treatment
Description: Complete Cell Cycle Arrest (CCCA): Ki-67 expression ≤ 2.7% after 14/28 days (+/- 2 days) of treatment.
  See general comments to biomarker endpoints above.
Time Frame: after 14/28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (20 missing in arm A; 41 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 160 | 138
Participants
  CCCA A1B2 = 0 (not achieved) | 160 | 138
  CCCA A1B2 = 1 (achieved) | 0 | 0
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.001, 95% CI 2-sided [-0.022 to 0.018] — [estimate comment as in outcome 8, analysis 1]

13. Secondary Outcome: Complete Cell Cycle Arrest (CCCA) After 28 Days (+/- 2 Days) of Treatment
Description: CCCA: Ki-67 expression ≤ 2.7%. Complete Cell Cycle Arrest (CCCA) defined as : Ki-67 ≤ 2.7%.
  See general comments to biomarker endpoints above.
Time Frame: after 28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (43 missing in arm A; 41 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 137 | 138
Participants
  CCCA A3B2 = 0 (not achieved) | 136 | 138
  CCCA A3B2 = 1 (achieved) | 1 | 0
Statistical Analysis 1: Comparison: Arm A; Test type: Superiority; Risk Difference (RD) = 0.007, 95% CI 2-sided [-0.017 to 0.034] — [estimate comment as in outcome 8, analysis 1]

14. Secondary Outcome: Low Cellularity (< 500 Tumor Cells) After 14 (Arm A)/28 Days (Arm B) (+/- 2 Days) of Treatment
Description: Low cellularity: < 500 tumor cells after 14/28 days (+/- 2 days) of treatment. See general comments to biomarker endpoints above.
Time Frame: after 14/28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (20 missing in arm A; 37 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 160 | 142
Participants
  Low Cell. A1B2 = 0 (not achieved) | 152 | 102
  Low Cell. A1B2 = 1 (achieved) | 8 | 40
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.229, 95% CI 2-sided [-0.31 to -0.148]; CI given as High posterior density interval (Bayesian confidence interval based on posterior distribution of effect/parameter of interest)

15. Secondary Outcome: Low Cellularity (< 500 Tumor Cells) After 28 Days (+/- 2 Days) of Treatment
Description: Low cellularity: < 500 tumor cells after 28 days (+/- 2 days) of treatment. See general comments to biomarker endpoints above.
Time Frame: after 28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (41 missing in arm A; 37 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 139 | 142
Participants
  Low Cell. A3B2 = 0 (not achieved) | 92 | 102
  Low Cell. A3B2 = 1 (achieved) | 47 | 40
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = 0.056, 95% CI 2-sided [-0.052 to 0.163] — [estimate comment as in outcome 8, analysis 1]

16. Secondary Outcome: Combined Early Response After 14 (Arm A)/28 (Arm B) Days (+/- 2 Days) of Treatment
Description: Combined early response defined by
  * CCCA (Ki-67 expression < 2.7%) or
  * low cellularity or
  * decrease of Ki-67 expression (versus baseline) by 30% or more or
  * TILs ≥ 60% See general comments to biomarker endpoints above.
Time Frame: after 14/28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (19 missing in arm A; 37 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 161 | 142
Participants
  Combined Resp. A1B2 = 0 (not achieved) | 116 | 53
  Combined Resp. A1B2 = 1 (achieved) | 45 | 89
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = -0.343, 95% CI 2-sided [-0.447 to -0.238]; [other analysis details as in outcome 14, analysis 1]

17. Secondary Outcome: Combined Early Response After 28 Days (+/- 2 Days) of Treatment
Description: as for outcome 16
Time Frame: after 28 days (+/- 2 days) of treatment
Population: Analyzed were all available samples of participants (41 missing in arm A; 37 missing in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 139 | 142
Participants
  Combined Resp. A3B2 = 0 (not achieved) | 47 | 53
  Combined Resp. A3B2 = 1 (achieved) | 92 | 89
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; Risk Difference (RD) = 0.035, 95% CI 2-sided [-0.076 to 0.146] — [estimate comment as in outcome 8, analysis 1]

18. Secondary Outcome: Disease Free Survival (DFS)
Description: Disease free survival (DFS) defined as time from the first date of no disease [i.e. date of surgery] to the first occurrence of disease recurrence or death from any cause.
Time Frame: from randomization up to 24 months until date of occurrence of no disease to the first occurrence of disease recurrence or death from any cause
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 180 | 179
Participants | 15 | 10
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.290, Regression, Cox; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.69 to 3.43]

19. Secondary Outcome: Overall Survival (OS).
Description: Overall survival (OS) defined as length of time from randomization to death from any cause. Given that novel post-neoadjuvant treatment options (on and off-trial) have emerged such as Pembrolizumab, the post-neoadjuvant treatment in the follow-up phase of this study would have been most certainly highly heterogeneous. Thus, completion of follow-up to 3 years was no longer justified. Therefore, follow-up was limited to 2 years and only clinically significant survival signals were observed.
Time Frame: from randomization up to 24 months until date of death from any cause.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 180 | 179
Participants | 5 | 3
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.495, Regression, Cox; Hazard Ratio (HR) = 1.65, 95% CI 2-sided [0.39 to 6.89]

20. Secondary Outcome: Event Free Survival (EFS)
Description: Event free survival (EFS) defined as length of time after randomization till death from any cause, failure to achieve remission after induction therapy, relapse in any site, or second malignancy
Time Frame: from randomization up to 24 months until date of death from any cause, failure to achieve remission after induction therapy, relapse in any site, or second malignancy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 180 | 179
Participants | 20 | 16
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.529, Regression, Cox; Univariable Cox Regression; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.64 to 2.38]

ADVERSE EVENTS:
Time Frame: AEs were recorded until 30 days after the last dose of study treatment or until initiation of new anticancer therapy, whichever occured first; SAEs were reported until 90 days after the last dose of study treatment or until initiation of new anticancer therapy. Therefore, AEs were usually reported for 29 - 30 weeks for participants in Arm A and 27 - 28 weeks for participants in Arm B. Data for survival analyses (OS, PFS) were assessed from randomization up to 24 months.
Description: In accordance with the protocol and SAP, AEs and SAEs were only collected for the neoadjuvant therapy until surgery.
  Non-serious adverse events with a frequency between 5 and 10% were not included in the CSR. In order to comply with the reporting requirements of ClinicalTrials.gov, the data for this area was re-evaluated using a different analysis programme (SAS) due to organisational restructuring.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 1/180 | 0/179
Serious Adverse Events (participants affected / at risk) | 86/178 | 87/178
Other Adverse Events (participants affected / at risk) | 178/178 | 178/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=178) | Arm B (N=178)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 23 | 21
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 10
Pancytopenia (Blood and lymphatic system disorders) | 9 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Immune-mediated myocarditis (Cardiac disorders) | 0 | 1
Addison's disease (Endocrine disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Device related thrombosis (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 12 | 9
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 22 | 12
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 2
Drug hypersensitivity (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 2
Immune-mediated adverse reaction (Immune system disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 2 | 1
Coronavirus infection (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 3
Gastrointestinal infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 3 | 2
Influenza (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 2
Wound infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Medical observation (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Fine motor skill dysfunction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Meningism (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Central venous catheter removal (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=178) | Arm B (N=178)
Anaemia (Blood and lymphatic system disorders) | 93 | 108
Leukopenia (Blood and lymphatic system disorders) | 51 | 49
Neutropenia (Blood and lymphatic system disorders) | 106 | 98
Thrombocytopenia (Blood and lymphatic system disorders) | 66 | 66
Constipation (Gastrointestinal disorders) | 44 | 52
Diarrhoea (Gastrointestinal disorders) | 46 | 58
Dyspepsia (Gastrointestinal disorders) | 22 | 25
Nausea (Gastrointestinal disorders) | 91 | 99
Stomatitis (Gastrointestinal disorders) | 24 | 31
Vomiting (Gastrointestinal disorders) | 40 | 26
Fatigue (General disorders) | 98 | 105
Mucosal inflammation (General disorders) | 39 | 21
Pyrexia (General disorders) | 44 | 26
Alanine aminotransferase increased (Investigations) | 47 | 37
Aspartate aminotransferase increased (Investigations) | 35 | 21
Neutrophil count decreased (Investigations) | 38 | 47
Platelet count decreased (Investigations) | 19 | 33
White blood cell count decreased (Investigations) | 18 | 29
Decreased appetite (Metabolism and nutrition disorders) | 18 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 32
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 32
Dysgeusia (Nervous system disorders) | 16 | 20
Headache (Nervous system disorders) | 39 | 41
Peripheral sensory neuropathy (Nervous system disorders) | 29 | 25
Polyneuropathy (Nervous system disorders) | 43 | 50
Insomnia (Psychiatric disorders) | 20 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 37 | 31
Alopecia (Skin and subcutaneous tissue disorders) | 91 | 99
Dry skin (Skin and subcutaneous tissue disorders) | 19 | 22
Rash (Skin and subcutaneous tissue disorders) | 32 | 27
Hot flush (Vascular disorders) | 32 | 21
Tachycardia (Cardiac disorders) | 5 | 9
Vertigo (Ear and labyrinth disorders) | 13 | 17
Hyperthyroidism (Endocrine disorders) | 12 | 10
Hypothyroidism (Endocrine disorders) | 8 | 12
Dry eye (Eye disorders) | 11 | 8
Abdominal pain (Gastrointestinal disorders) | 7 | 11
Abdominal pain upper (Gastrointestinal disorders) | 17 | 11
Dysphagia (Gastrointestinal disorders) | 10 | 9
Oral pain (General disorders) | 9 | 5
Chills (General disorders) | 14 | 10
Influenza like illness (General disorders) | 10 | 5
Mucosal dryness (General disorders) | 9 | 11
Oedema (General disorders) | 5 | 13
Oedema peripheral (General disorders) | 10 | 11
Hepatotoxicity (Hepatobiliary disorders) | 16 | 11
Drug hypersensitivity (Immune system disorders) | 11 | 8
Hypersensitivity (Immune system disorders) | 9 | 7
Cystitis (Infections and infestations) | 11 | 4
Urinary tract infection (Infections and infestations) | 11 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 14 | 13
Blood alkaline phosphatase increased (Investigations) | 8 | 11
Gamma-glutamyltransferase increased (Investigations) | 12 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8
Dizziness (Nervous system disorders) | 11 | 10
Paraesthesia (Nervous system disorders) | 8 | 11
Taste disorder (Nervous system disorders) | 14 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 15
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Erythema (Skin and subcutaneous tissue disorders) | 9 | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 11 | 6
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 9
Skin toxicity (Skin and subcutaneous tissue disorders) | 8 | 9

LIMITATIONS AND CAVEATS:
Although the trial had to stop recruitment prematurely after a first planned interim analysis of the first 100 pCR results (given that a probability of less than 2.5% of meeting the primary endpoint was estimated), 442 patients had already been screened and 363 had been randomized and were allowed to continue therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04770272/Prot_SAP_000.pdf